CLINICAL TRIAL: NCT04013763
Title: Outcome of Specific IgE Level in Children With IgE-mediated Wheat Allergy After Stop Using Wheat Containing Skin Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 1. Limit number of patients during COVID-19 situation
  2. Too small number of wheat allergic patients who are using wheat containing soap
Sponsor: Mahidol University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 038/2562(EC1)
Record Dates: First submitted 2019-07-01; First posted 2019-07-10 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Wheat Allergy; Children
Keywords: wheat allergy; skin sensitization; specific IgE; wheat containing skin care
MeSH Terms: conditions — Wheat Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Atopic dermatitis with stop using product (Experimental): case wheat allergy with atopic dermatitis and stop using wheat containing skin care products
  Interventions: Other: wheat containing skin care products
- Atopic dermatitis with containing using product (Experimental): case wheat allergy with atopic dermatitis and continue using wheat containing skin care products
  Interventions: Other: wheat containing skin care products
- Non atopic dermatitis with stop using product (Experimental): case wheat allergy with normal skin and stop using wheat containing skin care products
  Interventions: Other: wheat containing skin care products
- Non atopic dermatitis with continue using product (Experimental): case wheat allergy with normal skin and continue using wheat containing skin care products
  Interventions: Other: wheat containing skin care products
- Atopic dermatitis with no product use (No Intervention): case wheat allergy who does not use wheat containing skin care products and has atopic dermatitis
- Non atopic dermatitis with no product use (No Intervention): case wheat allergy who does not use wheat containing skin care products and no atopic dermatitis

INTERVENTIONS:
Other: wheat containing skin care products — stop or continue using wheat containing skin care products
  Arms: Atopic dermatitis with containing using product; Atopic dermatitis with stop using product; Non atopic dermatitis with continue using product; Non atopic dermatitis with stop using product

SUMMARY:
Wheat allergy is increasing in Thailand. Some studies show that cutaneous exposure of allergen may cause allergy and there are many wheat containing skin care products that are over-the-counter. So the purpose of our study is to determine level of specific immunoglobulin E antibodies to wheat and omega-5 gliadin in wheat allergy patients after stop using wheat containing skin care products.

DETAILED DESCRIPTION:
All children in this study were sensitized to wheat. Each patient was clinically evaluated, with focus on wheat allergy by medical history, medical examination included skin status (suspected atopic dermatitis or not). Blood sample was taken for baseline determination of immunoglobulin E antibodies to wheat and to omega-5 gliadin. Transepidermal water loss was examined in case with atopic dermatitis. The primary outcome was the specific immunoglobulin E antibodies to wheat and omega-5 gliadin in case that stop using wheat containing skin care product and case that continue using products.

ELIGIBILITY:
Inclusion Criteria:

* children age 1 to 18 years
* History of IgE-mediated wheat allergy

Exclusion Criteria:

* Parents refused to sign the consent
* severe atopic dermatitis
* on oral immunothery
* severe IgE mediated reaction after using wheat containing skin care product

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Specific IgE to wheat and omega-5 gliadin level | 1 year
  To follow-up the level of wheat and omega5 gliadin specificIgE after stop using the wheat containing skin care product compare to patients who continue using the product.

SECONDARY OUTCOMES:
level of transepidermal water loss | 1 year
  To follow up the transepidermal water loss in patients with atopic dermatitis, comparing the group that continue using the product to the group that stop using the product.

CONTACTS AND LOCATIONS:
Overall Officials: Punchama Pacharn, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj hospital, Bangkok Noi, Bangkok, Thailand

REFERENCES:
- [Result] Nakamura M, Yagami A, Hara K, Sano A, Kobayashi T, Aihara M, Hide M, Chinuki Y, Morita E, Teshima R, Matsunaga K. A new reliable method for detecting specific IgE antibodies in the patients with immediate type wheat allergy due to hydrolyzed wheat protein: correlation of its titer and clinical severity. Allergol Int. 2014 Jun;63(2):243-9. doi: 10.2332/allergolint.13-OA-0618. Epub 2014 Apr 25. PMID 24759554